CLINICAL TRIAL: NCT03351972
Title: Does Bowel Preparation (Either as a Single or Divided Dose) Produce Better Cleansing and Diagnostic Yield Than no Preparation at All in Small Bowel Capsule Endoscopy
Brief Title: Differences in Preparation for Small Bowel Capsule Endoscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Hotel Dieu Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STH20061
Record Dates: First submitted 2017-11-17; First posted 2017-11-24 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Capsule Endoscopy; Inflammatory Bowel Diseases; Celiac Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Celiac Disease | interventions — klean prep; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bowel Prep routine (Active Comparator): Participants randomised to this arm will receive their bowel prep (Klean Prep) with the routine guidance of taking the contents the day before their capsule endoscopy
  Interventions: Drug: Klean Prep
- Bowel Prep Split (Active Comparator): Participants randomised to this arm will receive their bowel prep (Klean Prep) with the guidance stating to take the first dose the day before the capsule endoscopy and the second dose the morning of the capsule endoscopy
  Interventions: Drug: Klean Prep
- No bowel prep (Experimental): Participants randomised to this arm will be advised to drink clear liquids only ahead of their capsule endoscopy procedure
  Interventions: Other: Clear liquids only

INTERVENTIONS:
Drug: Klean Prep — Participants randomised to use polyethylene glycol will follow either routine guidance of taking the bowel prep the night before their capsule endoscopy or receive guidance that they should split their dose between the night before and the morning of the procedure
  Other Names: Polyethylene Glycol
  Arms: Bowel Prep Split; Bowel Prep routine
Other: Clear liquids only — Participants randomised to clear liquids only will receive guidance to only drink clear liquids before their procedure
  Arms: No bowel prep

SUMMARY:
The introduction of video capsule endoscopy in 2000 has provided a convenient and minimally invasive imaging method for the whole small bowel. Capsule Endoscopy is used to investigate a number of conditions such as obscure gastrointestinal bleeding, iron deficiency anaemia, inflammatory bowel disease, celiac disease, small bowel tumors, and hereditary polyposis syndromes. However, Capsule Endoscopy capsules are not able to suction fluid or wash the intestine, thus making it susceptible to decreased visualization quality and diagnostic yield due to dark intestinal contents or air bubbles. In order to determine the best method for bowel preparation before Capsule Endoscopy, this study seeks to determine in patients undergoing small intestine Capsule Endoscopy if split dose Polyethylene Glycol or single morning dose of Polyethylene Glycol have a benefit in Visualisation quality when compared to clear fluids only. A co-primary outcome will also be the diagnostic yield, as measured by the aggregate of all the active preparation groups compared to than clear fluids only group. Secondary outcome measures will include tolerance of preparations, cleanliness as assessed by a validated 4 point scale, distal small bowel visualization (the last 1/4 of small bowel examination by time) and small bowel transit time (measured as time from first duodenal image to first cecal image). Adult outpatients referred for small bowel video capsule endoscopy will be considered for the study and this will run in the clinical environment as per routine. Patients will have been referred for capsule endoscopy as per normal clinical practice so not additional procedure will take place. Patients will be randomly assigned to in a one to one fashion to one of three groups in order to explore whether bowel preparation (either as a single or divided dose) produce better cleansing and diagnostic yield than no preparation at all in small bowel capsule endoscopy.

DETAILED DESCRIPTION:
In order to determine the best method for bowel preparation before Capsule Endoscopy, this study seeks to determine in patients undergoing small intestine Capsule Endoscopy if split dose Polyethylene Glycol or single morning dose of Polyethylene Glycol have a benefit in Visualisation quality when compared to clear fluids only. A co-primary outcome will also be the diagnostic yield, as measured by the aggregate of all the active preparation groups compared to than clear fluids only group. Secondary outcome measures will include tolerance of preparations, cleanliness as assessed by a validated 4 point scale, distal small bowel visualization (the last 1/4 of small bowel examination by time) and small bowel transit time (measured as time from first duodenal image to first cecal image).

Group Assignment:

The groups will have some common instructions: all groups will be instructed to stop iron supplements five days prior to the exam. On the day prior to the exam, patients will be instructed to have a light breakfast and lunch, followed by only clear fluids. Over the day, patients will be encouraged to have at least two litres of clear fluids. On the day of the exam, 80 mg of oral simethicone will be given 10 minutes prior to the exam. The capsule will be ingested at 9:00am, after which fluids may be consumed 2 hours later, and solid food 4 hours later. Patients will be randomly assigned to in a one to one fashion to one of three groups using a central online randomization program. The groups for this project include:

A. Control: no additional instructions beyond those above will be given. B. Single dose Polyethylene Glycol: Patients will take 2 litre of Polyethylene Glycol at 6am the day of the exam.

C. Split dose Polyethylene Glycol: Patients will take 1 litre of Polyethylene Glycol at 7pm the evening prior to the exam and 1 litre at 6am the day of the exam.

Recruitment of patients will be performed from outpatient gastroenterology clinics at Sheffield Teaching Hospitals NHS Trust. After a request for Capsule Endoscopy from a referring physician, the patient will be contacted by telephone by one of the Capsule endoscopy nurse specialists (who are also involved in the study) as per normal practice. The study will be discussed, the procedure explained and a convenient date for the procedure will be agreed with the patient. The patient will be invited to meet with one of the research staff at a mutually agreed time in order to go through the study once more and provide written consent should they agree to participate. Should they wish to participate but would prefer to complete a postal consent form, this will be arranged. The procedure will be completed according to normal practice. Patients will be advised that they can withdraw from the study at any point and choose a preferred option for bowel preparation

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients (18 years or older)
* routinely referred for small bowel video capsule endoscopy (CE)

Exclusion Criteria:

* dysphagia
* severe gastroparesis requiring endoscopic placement of capsule
* small bowel obstruction
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2017-11-23 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinician assessed Visual Quality of small bowel | 1 day
  Visual quality of the small bowel during capsule endoscopy as assessed by a clinician
clinician assessed Diagnostic yield during capsule endoscopy | 1 day
  Ability to produce a diagnosis following capsule endoscopy as assessed by a clinician

CONTACTS AND LOCATIONS:
Overall Officials: Mark McAlindon, MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (2):
- Hotel Dieu Hospital, Kingston, Ontario, Canada
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The study has been set-up and designed to ensure no IPD is shared